CLINICAL TRIAL: NCT00768053
Title: Open-Label Study To Evaluate The EULAR-RAID Score, Rheumatoid Arthritis Impact Of Disease Score, In Rheumatoid Arthritis Patients Eligible To Etanercept And Who Will Receive Etanercept
Brief Title: Evaluation of EULAR-RAID Score in Rheumatoid Arthritis Patients
Acronym: Rainbow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Lincoln Medical and Mental Health Center (Other); Umanis (Industry); SODIA (Unknown); depolabo (Unknown)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0881X1-4508; B1801019
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis
Keywords: EULAR-RAID; active rheumatoid arthritis; etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg once a week

SUMMARY:
The Disease Activity Score (DAS) is a system of measurement developed in the 1980s that uses certain criteria, including joint counts and patient perceived disease activity, to measure disease activity in people with Rheumatoid Arthritis . More recently, the European League against Rheumatism (EULAR) has developed a new system of measurement known as the Rheumatoid Arthritis Impact of Disease score, or EULAR-RAID score. The EULAR-RAID score is a composite score based on patient reported outcomes, and includes such criteria as pain, functional disability, fatigue, sleep disturbances, coping, overall assessment of physical well being and overall assessment of psychological well being. The objective of this study is to evaluate the practical modalities and performance of the EULAR- RAID score in patients with rheumatoid arthritis who have been prescribed etanercept as part of usual medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged up to or equal 18 years
* Meet the 1987 ACR Revised Criteria for Rheumatoid Arthritis.
* Active rheumatoid arthritis with a DAS greater than 3,2 and one of the two followings : Objective evidence of 4 clinical synovitis or CRP (plasma C-reactive protein) greater than 10 mg/l or ESR (erythrocyte sedimentation rate) greater than 28 mm/h
* Failure of MTX, taken for at least 3 months and at least 15 mg/wk or maximal tolerated dosage . In patients with contraindications or intolerance to MTX, failure of another drug with structural efficacy (leflunomide or sulfasalazine), taken for at least 3 months at the optimal tolerated dosage Concomitant treatment for RA : DMARDs, corticosteroids, NSAIDs and analgesics are permitted. DMARDs and corticosteroids should be stable between screening and baseline visits.
* Functional status Class I, II or III as defined by American College of Rheumatology (ACR) Revised Criteria.
* Negative serum beta-human chorionic gonadotropin (beta-HCG) pregnancy test at screening for all women of childbearing potential. Sexually active women of childbearing potential must use a medically acceptable form of contraception. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception. Sexually active men must agree to use a medically accepted form of contraception during the study.
* Able and willing to self-inject ETN or have a designee who can do so.
* Able to store injectable test article at 2 Celcius degree to 8 Celcius degree

Exclusion Criteria:

* Prior experience of biologic treatment for their RA including ETN.
* Sepsis or risk of sepsis.
* Current or recent infections, including chronic or localized.
* Planned orthopedic surgery within 3 months (for RA disease)
* History of orthopedic surgery 1 month before screening
* Latex sensitivity.
* Vaccination with live vaccine in the last 4 weeks, or expected to require such vaccination during the course of the study.
* Previous clinical trial involvement in the last 3 months.
* Patients with the following conditions or risk factors should only be entered into the study if the investigator has conducted and documented a full risk/benefit evaluation
* History of recurring or chronic infection, or underlying condition which may predispose patients to infections e.g. tuberculosis (TB) infection (Note: follow SmPC and French guidelines for appropriate screening and treatment of TB in the setting of anti-tumor necrosis factor (anti-TNF) therapy. Patients with latent TB (contact with TB patients, history of primary TB, intradermal test with 5 IU of tuberculin greater than 5 mm, or radiographic lung density greater than 1 cm and consistent with TB) should receive appropriate prophylactic therapy as recommended by the French Agency for healthcare Product Safety (AFSSAPS, http//afassaps.sante.fr/), serious infection (infection associated with hospitalization and/or intravenous antibiotics) within 1 month of test article administration or active infection at screening, open cutaneous ulcers, known human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) positive.
* Current or prior history of blood dyscrasias. Abnormal safety baseline blood test e.g. hemoglobin <= 85 g/L; hematocrit less than 27 %; platelet count less than 125 x 109/L; white blood cell count less than 3.5 x 109/L; serum creatinine greater than 175 µmol/L; aspartate aminotransferase (AST [SGOT]) and alanine aminotransferase (ALT [SGPT]) greater than 2 times the laboratory's upper limit of normal.
* Pre-existing or recent onset central nervous system (CNS) demyelinating disease.
* Cardiovascular conditions, e.g., myocardial infarction within 12 months of the screening visit, unstable angina pectoris, class III or IV congestive heart failure as defined by the New York Heart Association classification or decompensated congestive heart failure.
* Uncontrolled conditions, e.g., diabetes mellitus, hypertension (defined as screening systolic blood pressure greater than 160 mm Hg or screening diastolic blood pressure greater than 100 mm Hg), severe pulmonary disease requiring hospitalization or supplemental oxygen.
* At increased risk of malignancy.
* Reasonable expectation that the subject will not be able to satisfactorily complete the study.
* History of or current psychiatric illness, alcohol or drug abuse that would interfere with the subject's ability to comply with protocol requirements or give informed consent.
* Employment by the investigator or reporting directly or indirectly to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- France (15):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Belfort
  - Pfizer Investigational Site, Berck
  - Pfizer Investigational Site, Bonneville
  - Pfizer Investigational Site, Cahors
  - Pfizer Investigational Site, Corbeil-Essonnes
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Lomme
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rodez
  - Pfizer Investigational Site, Saint-Priest-en-Jarez
  - Pfizer Investigational Site, Valenciennes
- Pfizer Investigational Site, Monaco, Monaco

REFERENCES:
- [Derived] Duarte C, Santos EJF, Ferreira RJO, Kvien TK, Dougados M, de Wit M, da Silva JAP, Gossec L. Validity and reliability of the EULAR instrument RAID.7 as a tool to assess individual domains of impact of disease in rheumatoid arthritis: a cross-sectional study of 671 patients. RMD Open. 2021 Feb;7(1):e001539. doi: 10.1136/rmdopen-2020-001539. PMID 33547229
- [Derived] Dougados M, Brault Y, Logeart I, van der Heijde D, Gossec L, Kvien T. Defining cut-off values for disease activity states and improvement scores for patient-reported outcomes: the example of the Rheumatoid Arthritis Impact of Disease (RAID). Arthritis Res Ther. 2012 May 30;14(3):R129. doi: 10.1186/ar3859. PMID 22647431
- [Derived] Dougados M, Ripert M, Hilliquin P, Brocq O, Brault Y, Logeart I. Onset of action of etanercept in rheumatoid arthritis based on patient-reported outcomes. Clin Exp Rheumatol. 2012 Mar-Apr;30(2):266-8. Epub 2012 Apr 13. PMID 22325048
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4508&StudyName=Evaluation%20of%20EULAR-RAID%20score%20in%20Rheumatoid%20Arthritis%20patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study duration includes a screening period of up to 6 weeks, a 12 week open-label treatment period, and a 4 week follow-up period (telephone contact for the assessment of adverse events).
Groups:
- Etanercept (ETN): Subcutaneous (sc) injection once weekly using the 50 milligram (mg) pre-filled syringe during the 12-week treatment phase.
Period: Overall Study
Arm/Group | Etanercept (ETN)
Started | 108
Completed | 97
Not Completed | 11
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
Age Continuous [Mean (Standard Deviation); unit: years] | 53.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Reliability of the European League Against Rheumatism - Rheumatism Arthritis Impact of Disease (EULAR-RAID) Score
Description: EULAR-RAID score reliability assessed using an intraclass correlation coefficient (using a consistency definition where the between-measure variance is excluded from the denominator variance and its 95% confidence interval) and the standard error of measurement (SEM) and its 95% confidence interval (CI). A higher intraclass correlation coefficient (ICC) indicates greater score reliability (0.0 to 0.10=virtually none; 0.11 to 0.40=slight; 0.41 to 0.60=fair; 0.61 to 0.80=moderate; 0.81 to 1.00=substantial).
Time Frame: Screening, baseline
Population: All injected subjects population: received at least 1 dose of study treatment (same as Safety population).
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
intraclass correlation coefficient | 0.85 [0.79 to 0.90]
Statistical Analysis 1: Comparison: Etanercept (ETN); Intraclass correlation coefficient (ICC); Test type: Superiority or Other; p = 0.000, F test — F test for H0: ICC = 0
Statistical Analysis 2: Comparison: Etanercept (ETN); Standardized response mean: standard error of measurement; Test type: Superiority or Other; standard error of measurement = 0.65, 95% CI 2-sided [0.57 to 0.75]

2. Primary Outcome: Simplicity: Time for Completion of the EULAR-RAID Questionnaire
Description: EULAR-RAID is an assessment of patient reported outcomes for pain, functional disability, fatigue, sleep disturbance, coping, overall assessments of physical well-being and emotional well-being based on 7 numerical rating scales (NRS) questions. NRS individual questions with range of 0 (not affected, very good) to 10 (most affected) weighted and calculated with a total score range of 0 (not affected, very good) to 10 (most affected).
Time Frame: Baseline up to Week 12
Population: All injected subjects population. Data was not summarized; the time to complete the EULAR-RAID questionnaire was not analyzed separately from other components of the EULAR questionnaire (EULAR-RAID, questions on pain, Modified Health Assessment Questionnaire, sleep and coping)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 0

3. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Disease Activity Score Based on 28-joints Count (DAS28)
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity question measured on an 11-point rating scale scored 0 [none] to 10 [extreme]). Face validity assessed using a correlation coefficient between the EULAR-RAID score and the DAS28. A higher correlation coefficient indicates greater EULAR-RAID score validity.
Time Frame: Baseline, Week 4
Population: All injected subjects population
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient
  Baseline | 0.33 [0.15 to 0.49]
  Week 4 | 0.64 [0.50 to 0.74]
Statistical Analysis 1: Comparison: Etanercept (ETN); Week 4; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

4. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Disease Activity Score Based on 28-joints Count (DAS28): Week 12
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, ESR (mm/hour) and patient's global assessment of disease activity (participant rated arthritis activity question measured on an 11-point rating scale scored 0 [none] to 10 [extreme]). Face validity assessed using a correlation coefficient between the EULAR-RAID score and the DAS28. A higher correlation coefficient indicates greater EULAR-RAID score validity.
Time Frame: Week 12
Population: All injected subjects population
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient | 0.55 [0.40 to 0.68]
Statistical Analysis 1: Comparison: Etanercept (ETN); Week 12; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

5. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Disease Activity Score Based on 28-joints Count (DAS28): Time-normalized Average
Description: Time-normalized average is the area under the curve (AUC) / time between first and last observations. DAS28 calculated from number of swollen joints and painful joints using 28 joints count, ESR (mm/hour) and patient's global assessment of disease activity (participant rated arthritis activity question measured on an 11-point rating scale scored 0 [none] to 10 [extreme]). Face validity assessed using a correlation coefficient between the EULAR-RAID and DAS28 scores. A higher correlation coefficient indicates greater EULAR-RAID score validity.
Time Frame: Baseline, Last observation up to Week 12
Population: All injected subjects population; score profile from baseline to last observation post-baseline.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient | 0.59 [0.45 to 0.70]
Statistical Analysis 1: Comparison: Etanercept (ETN); Time-normalized average; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

6. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Patient Global Assessment (PGA) of Health Status
Description: PGA of health status is a single-item participant rated response to the question "in general, how would you rate your health over the last 2 to 3 weeks"; scored 0 (very well) to 10 (extremely bad). Face validity assessed using a correlation coefficient between the EULAR-RAID score and the PGA. A higher correlation coefficient indicates greater EULAR-RAID score validity (best >0.85).
Time Frame: Baseline, Week 4
Population: All injected subjects population
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient
  Baseline | 0.77 [0.68 to 0.84]
  Week 4 | 0.93 [0.90 to 0.95]
Statistical Analysis 1: Comparison: Etanercept (ETN); Week 4; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

7. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Patient Global Assessment (PGA) of Health Status: Week 12
Description: PGA of health status is a single-item participant rated response to the question "in general, how would you rate your health over the last 2 to 3 weeks"; scored 0 (very well) to 10 (extremely bad). Face validity assessed using a correlation coefficient between the EULAR-RAID score and PGA health status score. A higher correlation coefficient indicates greater EULAR-RAID score validity (best >0.85).
Time Frame: Week 12
Population: All injected subjects population
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient | 0.89 [0.84 to 0.93]
Statistical Analysis 1: Comparison: Etanercept (ETN); Week 12; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

8. Primary Outcome: Face Validity: Correlation Coefficients of the EULAR-RAID Score With the Patient Global Assessment (PGA) of Health Status: Time-normalized Average
Description: Time-normalized average is the area under the curve (AUC) / time between first and last observations. PGA of health status is a single-item participant rated response to the question "in general, how would you rate your health over the last 2 to 3 weeks"; scored 0 (very well) to 10 (extremely bad). Face validity assessed using a correlation coefficient between the EULAR-RAID score and PGA health status score. A higher correlation coefficient indicates greater EULAR-RAID score validity (best >0.85).
Time Frame: Baseline, Last observation up to Week 12
Population: All injected subjects population; score profile from baseline to last observation post-baseline.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
correlation coefficient | 0.92 [0.89 to 0.95]
Statistical Analysis 1: Comparison: Etanercept (ETN); Time-normalized average; Test type: Superiority or Other; p < 0.001, t-test for the Pearson correlation

9. Primary Outcome: Sensitivity to Change of the EULAR-RAID Score: Change From Baseline to Week 4
Description: Sensitivity to change analyzed by testing if the difference of change from baseline of EULAR-RAID score minus the change from baseline of each component (pain, functional disability, fatigue, sleep disturbance, coping, overall physical and emotional well-being with score range 0 [not affected, very good] to 10 [most affected]) was different from 0 or not. Results expressed as standardized response mean (SRM) calculated as ratio of mean change over standard deviation of the change. A non significant test (p value ≥0.05) means the component had a significant influence to global EULAR RAID score.
Time Frame: Baseline, Week 4
Population: All injected subjects population
Measure: Number; unit: standardized response mean
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
standardized response mean
  EULAR-RAID score | -1.01
  Pain NRS value | -1.06
  Functional disability NRS value | -1.02
  Fatigue NRS value | -0.86
  Sleep NRS value | -0.64
  Physical well-being NRS value | -0.90
  Emotional well-being NRS value | -0.68
  Coping NRS value | -0.60
Statistical Analysis 1: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Pain NRS value; Test type: Superiority or Other; p < 0.001, paired t-test; A non significant test (p-value ≥ 0.05) would indicate the component had a significant influence to the global EULAR-RAID score
Statistical Analysis 2: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Functional disability NRS value; Test type: Superiority or Other; p < 0.001, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Fatigue NRS value; Test type: Superiority or Other; p = 0.837, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Sleep NRS value; Test type: Superiority or Other; p = 0.035, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Physical well-being NRS value; Test type: Superiority or Other; p = 0.351, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Emotional well-being NRS value; Test type: Superiority or Other; p = 0.025, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Coping NRS value; Test type: Superiority or Other; p < 0.001, paired t-test; [statistical method as in outcome 9, analysis 1]

10. Primary Outcome: Sensitivity to Change of the EULAR-RAID Score: Change From Baseline to Week 12
Description: as for outcome 9
Time Frame: Baseline, Week 12
Population: All injected subjects population
Measure: Number; unit: standardized response mean
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
standardized response mean
  EULAR-RAID score | -1.37
  Pain NRS value | -1.37
  Functional disability NRS value | -1.24
  Fatigue NRS value | -1.15
  Sleep NRS value | -0.92
  Physical well-being NRS value | -1.27
  Emotional well-being NRS value | -1.06
  Coping NRS value | -0.96
Statistical Analysis 1: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Pain NRS value; Test type: Superiority or Other; p < 0.001, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Functional disability NRS value; Test type: Superiority or Other; p = 0.052, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Fatigue NRS value; Test type: Superiority or Other; p = 0.895, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Sleep NRS value; Test type: Superiority or Other; p = 0.153, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Physical well-being NRS value; Test type: Superiority or Other; p = 0.029, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Emotional well-being NRS value; Test type: Superiority or Other; p = 0.043, paired t-test; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Etanercept (ETN); Comparison of change from baseline between EULAR-RAID score and Coping NRS value; Test type: Superiority or Other; p < 0.001, paired t-test; [statistical method as in outcome 9, analysis 1]

11. Secondary Outcome: Percentage of Participants Achieving a Moderate or Good EULAR Response Rate at Week 12
Description: EULAR response rate is based on DAS28. For DAS28 ≤3.2 at observation (low disease activity), change from baseline of <-1.2=good response or ≥-1.2 to <-0.6=moderate response; DAS28 >3.2 to 5.1 at observation (moderate or high disease activity), change from baseline of <-1.2 or ≥-1.2 to <-0.6=moderate response; DAS28 >5.1 (high disease activity) at observation, change from baseline of <-1.2=moderate response. DAS28 calculated using the 28 joints count, ESR mm/hour, and PGA of disease activity (participant rated arthritis activity measured on 11-point rating scale: 0 [none] to 10 [extreme]).
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 95
percentage of participants | 87.4

12. Secondary Outcome: Minimal Clinically Important Improvement (MCII) of the EULAR-RAID Score: 75th Percentile of Change at Week 4 and Week 12
Description: MCII is a 2-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours. Question 1: in comparison to study start (Improved, No Change, or Worse). Question 2: if response was Improved, participant rated how important the improvement was (Very important, Moderately important, Slightly important, or Not important at all). The MCII score is defined as the 75th percentile of the change in EULAR-RAID score between baseline and observation among participants whose evaluation of the response therapy at observation was Moderately or Slightly important improvement.
Time Frame: Week 4, Week 12
Population: All injects subjects population; (n) includes participants with analyzable data at observation (responses of Yes or No).
Measure: Number; unit: scores on a scale
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
scores on a scale
  Week 4 (n=102) | -0.19
  Week 12 (n=99) | -1.29

13. Secondary Outcome: Percentage of Participants Achieving a Minimal Clinically Important Improvement (MCII) Score at Week 4 Who Had Moderately or Slightly Important Improvement at Week 4, Week 12, or Last Observation (Last Obs)
Description: MCII is a 2-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours. Question 1: in comparison to study start (Improved, No change, or Worse). Question 2: if response was Improved, participant rated how important the improvement was (Very important, Moderately important, Slightly important, or Not important at all). MCII score at Week 4 calculated on participants with Moderately or Slightly important improvement (Mod/Slightly Imp Improvement) achieved at observation.
Time Frame: Week 4, Week 12, and Last observation up to Week 12
Population: All injected subjects population; (n) includes participants with analyzable data at observation (responses of Yes or No).
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
percentage of participants
  Mod/Slightly Imp Improvement Week 4 (n=102) | 78.4
  Mod/Slightly Imp Improvement Week 12 (n=99) | 87.9
  Mod/Slightly Imp Improvement Last Obs (n=108) | 87.0

14. Secondary Outcome: Percentage of Participants Achieving a Minimal Clinically Important Improvement Score at Week 12 Who Had Moderately or Slightly Important Improvement at Week 4, Week 12, or Last Observation (Last Obs)
Description: MCII is a 2-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours. Question 1: in comparison to study start (Improved, No change, or Worse). Question 2: if response was Improved, participant rated how important the improvement was (Very important, Moderately important, Slightly important, or Not important at all). MCII score at Week 12 calculated on participants with Moderately or Slightly important improvement (Mod/Slightly Imp Improvement) achieved at observation.
Time Frame: Week 4, Week 12, and Last observation up to Week 12
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
percentage of participants
  Mod/Slightly Imp Improvement Week 4 (n=102) | 61.8
  Mod/Slightly Imp Improvement Week 12 (n=99) | 78.8
  Mod/Slightly Imp Improvement Last Obs (n=108) | 76.9

15. Secondary Outcome: Patient Acceptable Symptom State (PASS) of the EULAR-RAID Score: 75th Percentile of Change at Week 4 and Week 12
Description: PASS is a 1-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours (If you were to remain in the next few months as you were during the last hours, would this be Acceptable or Unacceptable to you?). PASS score is defined as the 75th percentile of the change in EULAR-RAID score between baseline and observation among participants whose evaluation of their symptom state at observation was Acceptable.
Time Frame: Week 4, Week 12
Population: All injected subjects population. Unacceptable value put to participants prematurely withdrawn or with missing data; (n) includes participants with analyzable data at observation (responses of Acceptable or Unacceptable).
Measure: Number; unit: scores on a scale
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
scores on a scale
  Week 4 (n=102) | 4.15
  Week 12 (=99) | 3.27

16. Secondary Outcome: Percentage of Participants Achieving a Patient Acceptable Symptom State (PASS) Score at Week 4 Who Had an Acceptable Symptom State at Week 4, Week 12, or Last Observation (Last Obs)
Description: PASS is a 1-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours (If you were to remain in the next few months as you were during the last hours, would this be acceptable or unacceptable to you?). PASS score at Week 4 calculated on participants with Acceptable symptom state achieved at observation.
Time Frame: Week 4, Week 12, and Last observation up to Week 12
Population: All injected subjects population; (n) includes participants with analyzable data at observation (responses of Acceptable or Unacceptable).
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
percentage of participants
  Acceptable Week 4 (n=102) | 57.8
  Acceptable Week 12 (n=99) | 74.7
  Acceptable Last Obs (n=108) | 72.2

17. Secondary Outcome: Percentage of Participants Achieving a Patient Acceptable Symptom State (PASS) Score at Week 12 Who Had an Acceptable Symptom State at Week 4, Week 12, or Last Observation (Last Obs)
Description: PASS is a 1-question assessment of how rheumatoid arthritis has affected the participant in the last 48 hours (If you were to remain in the next few months as you were during the last hours, would this be acceptable or unacceptable to you?). PASS score at Week 12 calculated on participants with Acceptable symptom state achieved at observation.
Time Frame: Week 4, Week 12, and Last observation up to Week 12
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 108
percentage of participants
  Acceptable Week 4 (n=102) | 49.0
  Acceptable Week 12 (n=99) | 64.6
  Acceptable Last Obs (n=108) | 62.0

18. Secondary Outcome: Percentage of Participants Achieving > 1.2 Improvement in DAS28 at Week 12
Description: DAS28 calculated from number of painful and swollen joints using 28 joints count (PJC, SJC), ESR (mm/hour), and patient's global assessment of disease activity (arthritis activity measured on 11-point rating scale scored 0 [none] to 10 [extreme]). DAS28 score calculated as 0.56*square root (√) (PJC28) + 0.28 *√ (SJC28) + 0.70*ln ESR + 0.014*PGA*10. DAS28 score >5.1=higher disease activity; ≤3.2=low disease activity; <2.6=clinical remission. Achievement of >1.2 improvement defined as decrease in DAS28 >1.2 (i.e., change in DAS28 < -1.2).
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 95
percentage of participants | 77.9

19. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 <2.6) at Week 12
Description: DAS28 calculated from number of painful and swollen joints using 28 joints count (PJC, SJC), ESR (mm/hour), and patient's global assessment of disease activity (arthritis activity measured on 11-point rating scalescored 0 [none] to 10 [extreme]). DAS28 score calculated as 0.56*square root (√) (PJC28) + 0.28 *√ (SJC28) + 0.70*ln ESR + 0.014*PGA*10. DAS28 score >5.1=higher disease activity; ≤3.2=low disease activity; <2.6=clinical remission.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 96
percentage of participants | 28.1

20. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (DAS28 ≤3.2) at Week 12
Description: DAS28 calculated from number of painful and swollen joints using 28 joints count (PJC, SJC), ESR (mm/hour), and patient's global assessment of disease activity (arthritis activity measured on 11-point rating scale scored 0 [none] to 10 [extreme]). DAS28 score calculated as 0.56*square root (√) (PJC28) + 0.28 *√ (SJC28) + 0.70*ln ESR + 0.014*PGA*10. DAS28 score >5.1=higher disease activity; ≤3.2=low disease activity; <2.6=clinical remission.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 96
percentage of participants | 46.9

21. Secondary Outcome: Percentage of Participants Achieving > 0.6 DAS28 Response at Week 12
Description: DAS28 calculated from number of painful and swollen joints using 28 joints count (PJC, SJC), ESR (mm/hour), and patient's global assessment of disease activity (arthritis activity measured on 11-point rating scale scored 0 [none] to 10 [extreme]). DAS28 score calculated as 0.56*square root (√) (PJC28) + 0.28 *√ (SJC28) + 0.70*ln ESR + 0.014*PGA*10. DAS28 score >5.1=higher disease activity; ≤3.2=low disease activity; <2.6=clinical remission. Achievement of >0.6 DAS28 response defined as decrease in DAS28 > 0.6 (i.e. change in DAS28 < -0.6).
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 95
percentage of participants | 91.6

22. Secondary Outcome: Time to Achievement of Sustained Low Disease Activity Score (LDAS): DAS28 ≤3.2
Description: Time to sustained LDAS measured as maintenance of low disease activity score beyond Week 12. DAS28 calculated from number of painful and swollen joints using 28 joints count (PJC, SJC), ESR (mm/hour), and patient's global assessment of disease activity (arthritis activity measured on 11-point rating scale scored 0 [none] to 10 [extreme]). DAS28 score calculated as 0.56*square root (√) (PJC28) + 0.28 *√ (SJC28) + 0.70*ln ESR + 0.014*PGA*10. DAS28 score >5.1=higher disease activity; ≤3.2=low disease activity; <2.6=clinical remission.
Time Frame: Baseline up to Week 12
Population: All injected subjects population; DAS28 assessed at Week 4 and Week 12; sustained LDAS could only have been observed beyond Week 12. Time to event analysis not possible within study duration.
Measure: Number; unit: participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 0

23. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Week 12
Description: American College of Rheumatology 20% (ACR20) response: responder = ≥20% improvement in tender and swollen joint count and ≥20% improvement in at least 3 of 5 ACR core measures: patient assessment of pain (scored 1=extreme pain to 6=no pain; score transformed to 0 to 100: higher score indicates less pain), Patient's Global Assessment and Physician's Global Assessment of disease activity (assess arthritis activity; both scored 0=none to 10=extreme), Modified Health Assessment Questionnaire (assess amount of difficulty to perform an activity scored 0=no difficulty to 3=unable to do), and ESR.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 94
percentage of participants | 71.3

24. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Week 12
Description: American College of Rheumatology 50% (ACR50) response: responder = ≥50% improvement in tender and swollen joint count and ≥50% improvement in at least 3 of 5 ACR core measures: patient assessment of pain (scored 1=extreme pain to 6=no pain; score transformed to 0 to 100: higher score indicates less pain), Patient's Global Assessment and Physician's Global Assessment of disease activity (assess arthritis activity; both scored 0=none to 10=extreme), Modified Health Assessment Questionnaire (assess amount of difficulty to perform an activity scored 0=no difficulty to 3=unable to do), and ESR.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 93
percentage of participants | 47.3

25. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70 Response at Week 12
Description: American College of Rheumatology 70% (ACR70) response: responder = ≥70% improvement in tender and swollen joint count and ≥70% improvement in at least 3 of 5 ACR core measures: patient assessment of pain (scored 1=extreme pain to 6=no pain; score transformed to 0 to 100: higher score indicates less pain), Patient's Global Assessment and Physician's Global Assessment of disease activity (assess arthritis activity; both scored 0=none to 10=extreme), Modified Health Assessment Questionnaire (assess amount of difficulty to perform an activity scored 0=no difficulty to 3=unable to do), and ESR.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 98
percentage of participants | 16.3

26. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 90 Response at Week 12
Description: American College of Rheumatology 90% (ACR90) response: responder = ≥90% improvement in tender and swollen joint count and ≥90% improvement in at least 3 of 5 ACR core measures: patient assessment of pain (scored 1=extreme pain to 6=no pain; score transformed to 0 to 100: higher score indicates less pain), Patient's Global Assessment and Physician's Global Assessment of disease activity (assess arthritis activity; both scored 0=none to 10=extreme), Modified Health Assessment Questionnaire (assess amount of difficulty to perform an activity scored 0=no difficulty to 3=unable to do), and ESR.
Time Frame: Week 12
Population: All injected subjects population; N=number of participants with evaluable data at observation.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept (ETN)
Number analyzed (Participants) | 99
percentage of participants | 3.0

ADVERSE EVENTS:
Time Frame: Time the Informed Consent Form was signed up to Week 16 Follow-up visit
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept (ETN)
Serious Adverse Events (participants affected / at risk) | 5/108
Other Adverse Events (participants affected / at risk) | 53/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (ETN) (N=108)
Abdominal pain (Gastrointestinal disorders) | 1
Arthritis bacterial (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (ETN) (N=108)
Nausea (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 4
Fatigue (General disorders) | 4
Injection site erythema (General disorders) | 8
Injection site reaction (General disorders) | 18
Bronchitis (Infections and infestations) | 8
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Erythema (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.